CLINICAL TRIAL: NCT01244932
Title: Determination of the Minimum Effective Volume of Local Anesthetic Using Ultrasound Guidance for Interscalene Brachial Plexus Block
Brief Title: Minimum Effective Volume of Local Anesthetic Using Ultrasound for Brachial Plexus Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Luiz Fernando dos Reis Falcao, Ph.D., Federal University of São Paulo
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: UNIFESP-01
Record Dates: First submitted 2010-10-14; First posted 2010-11-22 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bupivacaine 0.5% — Patients will be given bupivacaine 0.5% in different doses (up-down study).

SUMMARY:
The purpose of this study is to determine the minimum effective volume of local anesthetic for interscalene brachial plexus block using ultrasound guidance and nerve stimulator guidance.

DETAILED DESCRIPTION:
This will be a single group assignment, double-blind, up-down sequential allocation study. Interscalene brachial plexus block (ISBPB) is a common nerve block given to patients who are undergoing shoulder surgery. This block has a low, but still significant, rate of complications. Reducing the volume of local anesthetic given during the block may allow some of these complications to be avoided. Participants will undergo ISBPB under ultrasound and nerve stimulator guidance. Patients will initially receive 15mL of local anesthetic (bupivacaine 0.5% with epinephrine). The volume used for each subsequent patient depends upon the success or failure of the previous patient's block - a failure will cause the volume given to increase by 1.0 mL, while a success will cause the volume to decrease by the same amount.

The goal of this study is to determine the minimum effective anesthetic volume of bupivacaine 0.5% providing anesthesia in patients when using ultrasound and nerve stimulator to guide placement of the block. The secondary outcome will be the evaluation of diaphragmatic function and post-surgery analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving interscalene brachial plexus block for shoulder surgery
* Age between 21 and 65 years
* ASA physical status I/II
* Body mass index < 35 kg/m2

Exclusion Criteria:

* Chronic obstructive pulmonary disease
* Psychiatric history
* Allergy to bupivacaine
* Infection in the site of block
* Coagulation disorders

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
ED95 of bupivacaine minimum effective volume | ED95
  The ED95 of bupivacaine minimum effective volume determination in interscalene brachial plexus block using ultrasound guidance. [ Time Frame: every 10 minutes until 30 minutes, after 4 hours and after 6 hours post-block ]

SECONDARY OUTCOMES:
Diaphragmatic Function | Diaphragmatic
  Diaphragmatic Function (as assessed by diaphragmatic movement on ultrasound) [ Time Frame: after 30 minutes, 4 hours and 6 hours post-block ]
Post-surgery analgesia | Analgesia
  Post-surgery analgesia [ Time Frame: after 4 hours and 6 hours post-block ]

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Fernando Falcao, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Luiz Fernando dos Reis Falcao, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Farquhar-Thomson DR, Baker AK, Satapathy AR, Coventry D, Harper GK, Stafford MA, Hill DA. Minimum volume of local anaesthetic required for an axillary brachial plexus block. Br J Anaesth. 2010 Sep;105(3):382-3. doi: 10.1093/bja/aeq220. No abstract available. PMID 20716568
- [Background] Ponrouch M, Bouic N, Bringuier S, Biboulet P, Choquet O, Kassim M, Bernard N, Capdevila X. Estimation and pharmacodynamic consequences of the minimum effective anesthetic volumes for median and ulnar nerve blocks: a randomized, double-blind, controlled comparison between ultrasound and nerve stimulation guidance. Anesth Analg. 2010 Oct;111(4):1059-64. doi: 10.1213/ANE.0b013e3181eb6372. Epub 2010 Aug 12. PMID 20705778
- [Background] Harper GK, Stafford MA, Hill DA. Minimum volume of local anaesthetic required to surround each of the constituent nerves of the axillary brachial plexus, using ultrasound guidance: a pilot study. Br J Anaesth. 2010 May;104(5):633-6. doi: 10.1093/bja/aeq050. Epub 2010 Mar 16. PMID 20233750
- [Background] Duggan E, El Beheiry H, Perlas A, Lupu M, Nuica A, Chan VW, Brull R. Minimum effective volume of local anesthetic for ultrasound-guided supraclavicular brachial plexus block. Reg Anesth Pain Med. 2009 May-Jun;34(3):215-8. doi: 10.1097/AAP.0b013e31819a9542. PMID 19587618
- [Background] O'Donnell BD, Iohom G. An estimation of the minimum effective anesthetic volume of 2% lidocaine in ultrasound-guided axillary brachial plexus block. Anesthesiology. 2009 Jul;111(1):25-9. doi: 10.1097/ALN.0b013e3181a915c7. PMID 19512869
- [Background] Gupta PK, Pace NL, Hopkins PM. Effect of body mass index on the ED50 volume of bupivacaine 0.5% for supraclavicular brachial plexus block. Br J Anaesth. 2010 Apr;104(4):490-5. doi: 10.1093/bja/aeq017. Epub 2010 Feb 18. PMID 20167584
- [Background] Marhofer P, Eichenberger U, Stockli S, Huber G, Kapral S, Curatolo M, Kettner S. Ultrasonographic guided axillary plexus blocks with low volumes of local anaesthetics: a crossover volunteer study. Anaesthesia. 2010 Mar;65(3):266-71. doi: 10.1111/j.1365-2044.2010.06247.x. Epub 2010 Jan 29. PMID 20121770
- [Background] Renes SH, Rettig HC, Gielen MJ, Wilder-Smith OH, van Geffen GJ. Ultrasound-guided low-dose interscalene brachial plexus block reduces the incidence of hemidiaphragmatic paresis. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):498-502. doi: 10.1097/AAP.0b013e3181b49256. PMID 19920426
- [Background] Smith HM, Duncan CM, Hebl JR. Clinical utility of low-volume ultrasound-guided interscalene blockade: contraindications reconsidered. J Ultrasound Med. 2009 Sep;28(9):1251-8. doi: 10.7863/jum.2009.28.9.1251. PMID 19710225
- [Derived] Falcao LF, Perez MV, de Castro I, Yamashita AM, Tardelli MA, Amaral JL. Minimum effective volume of 0.5% bupivacaine with epinephrine in ultrasound-guided interscalene brachial plexus block. Br J Anaesth. 2013 Mar;110(3):450-5. doi: 10.1093/bja/aes419. Epub 2012 Nov 29. PMID 23195326